CLINICAL TRIAL: NCT00896025
Title: A Multi-Center Trial to Study Acute Liver Failure: N-Acetylcysteine (NAC) Open Label Use Study
Brief Title: Study of N-Acetylcysteine in Acute Liver Failure (ALF)
Acronym: ONAC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This observational study was stopped after 140 patients were enrolled, no more funds available to continue.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012009-011; NIDDK U-01 058369
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Acute Liver Failure; Fulminant Hepatic Failure
Keywords: Liver disease
MeSH Terms: conditions — Liver Failure, Acute; Liver Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Open label-comparator is historical data.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetycylcysteine (Active Comparator): Each eligible Acute Liver Failure patient will be given N-acetylcysteine (NAC), beginning at a dose of 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour, followed by 50 mg/kg in 500 ml 5% dextrose over four hours, and 125 mg/kg in 1000 ml 5% dextrose over 19 hours, then 150 mg/kg in 1000 ml 5% dextrose per 24 hours for an additional 48 hours. The patient will be on continuous N-acetylcysteine infusion for a total of 72 hours.
  Interventions: Drug: N-acetylcysteine
- Standard of care (No Intervention): Each eligible Acute Liver Failure patient for whom the investigator chooses not to utilize N-acetylcysteine may serve as a control and receives standard of care.

INTERVENTIONS:
Drug: N-acetylcysteine — Patients will be included in the trial from the onset of any hepatic coma grade and will receive NAC for the following 72 hrs.
  NAC Solutions: The N-acetylcysteine will be added to 5% dextrose in defined concentrations according to the sequence of four specific doses required for the study.
  i.Solution A: 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour
  ii.Solution B: 50 mg/kg in 500 ml 5% dextrose over four hours
  iii.Solution C: 125 mg/kg in 1000 ml 5% dextrose over 19 hours
  iv.Solution D: 150 mg/kg in 1000 ml 5% dextrose per 24 hours
  v.Solution E: 150 mg/kg in 1000 ml 5% dextrose per 24 hours
  Other Names: Mucomyst
  Arms: N-acetycylcysteine

SUMMARY:
This proposed study is a multi-center open label study to determine if N-acetylcysteine has any survival benefits in patients with acute liver failure.

DETAILED DESCRIPTION:
Patients admitted to study sites with carefully defined criteria for acute liver failure and who are thought not to have acetaminophen toxicity, mushroom poisoning, pregnancy-related liver failure, or malignancy will be eligible. Each patient will receive intravenously in solution of 5% dextrose in water containing N-acetylcysteine, beginning at a dose of 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour, and in declining doses over a total of 72 hours. Care of patients and consideration of transplantation or other clinical decisions will not be affected by the study or the use of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent from patient's next of kin
* Altered mentation of any degree (encephalopathy)
* Evidence of moderately severe clotting abnormalities (international normalized ratio ≥ 1.5)
* A presumed acute illness onset of less than 26 weeks
* Admitted to study site hospital intensive care units with acute liver failure and who can be evaluated and started on treatment within the first 24 hours of hospitalization
* All subjects will be between 18 and 70 years
* The NIH guidelines on the inclusion of women and minorities as subjects will be observed

Exclusion Criteria:

* Patients less than age 18 or over 70 years of age
* Acetaminophen or mushroom poisoning induced liver failure
* Patients with a diagnosis of shock liver (ischemic hepatopathy)
* Acute liver failure of pregnancy
* Acute liver failure thought secondary to intra-hepatic malignancy
* Cerebral herniation
* Intractable arterial hypotension
* Severe sepsis (temperature >39º C and/or significant bacteremia) present at the time of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2008-12; Primary Completion 2015-10-15 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Lee, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Northwestern University Medical School, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital (Columbia and Cornel), New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stravitz RT, Fontana RJ, Karvellas C, Durkalski V, McGuire B, Rule JA, Tujios S, Lee WM; Acute Liver Failure Study Group. Future directions in acute liver failure. Hepatology. 2023 Oct 1;78(4):1266-1289. doi: 10.1097/HEP.0000000000000458. Epub 2023 May 16. PMID 37183883
- See also: Acute Liver Failure Website — http://www.acuteliverfailure.org

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetycylcysteine: Acute liver failure population
Period: Overall Study
Arm/Group | N-acetycylcysteine
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- N-acetycylcysteine: Each eligible Acute Liver Failure patient will be given N-acetylcysteine (NAC), beginning at a dose of 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour, followed by 50 mg/kg in 500 ml 5% dextrose over four hours, and 125 mg/kg in 1000 ml 5% dextrose over 19 hours, then 150 mg/kg in 1000 ml 5% dextrose per 24 hours for an additional 48 hours. The patient will be on continuous NAC infusion for a total of 72 hours.
Arm/Group | N-acetycylcysteine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 46 [23 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate With or Without Transplant
Description: The primary outcome is to compare all patients who survive (with or without transplant) to those who die.
Time Frame: 3 Weeks
Population: The estimated minimum enrollment for any statistical validity was 100 patients. Due to low enrollment (8 participants) and the likelihood of generating any meaningful study data moving forward, the DSMB recommended the early termination of the study. Data was not collected since study was terminated, therefore there was no data to analyze.
Groups:
- N-acetycylcysteine: Acute liver failure population
  N-acetylcysteine: Patients will be included in the trial from the onset of any hepatic coma grade and will receive NAC for the following 72 hrs.
  NAC Solutions: The N-acetylcysteine will be added to 5% dextrose in defined concentrations according to the sequence of four specific doses required for the study.
  i.Solution A: 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour
  ii.Solution B: 50 mg/kg in 500 ml 5% dextrose over four hours
  iii.Solution C: 125 mg/kg in 1000 ml 5% dextrose over 19 hours
  iv.Solution D: 150 mg/kg in 1000 ml 5% dextrose per 24 hours
  v.Solution E: 150 mg/kg in 1000 ml 5% dextrose per 24 hours
Arm/Group | N-acetycylcysteine
Number analyzed (Participants) | 0

2. Primary Outcome: Survival Rate With or Without Transplant
Description: The primary outcome is to compare all patients who survive (with or without transplant) to those who die.
Time Frame: 1-year follow-up
Population: The estimated minimum enrollment for any statistical validity was 100 patients. Due to low enrollment (8 participants) and the likelihood of generating any meaningful study data moving forward, the DSMB recommended the early termination of the study. Data was not collected since study was terminated.
Arm/Group | N-acetycylcysteine
Number analyzed (Participants) | 0

3. Primary Outcome: Survival Rate With or Without Transplant
Description: The primary outcome is to compare all patients who survive (with or without transplant) to those who die.
Time Frame: 2-year follow-up
Population: as for outcome 2
Arm/Group | N-acetycylcysteine
Number analyzed (Participants) | 0

4. Secondary Outcome: To Compare Patients Who Survive Without Transplantation to All Other Patients Enrolled in This Study (Those Who Receive a Transplant and Live, Those Who Receive a Transplant and Die, or Those Who Die Before Transplantation).
Description: The estimated minimum enrollment for any statistical validity was 100 patients. Due to low enrollment (8 participants) and the likelihood of generating any meaningful study data moving forward, the DSMB recommended the early termination of the study. Data was not collected since study was terminated, therefore no data to analyze.
Time Frame: 3 Week follow-up
Population: Data was not collected since study was terminated, therefore there was no data to analyze.
Groups:
- N-acetycylcysteine: Each eligible Acute Liver Failure patient will be given N-acetylcysteine (NAC), beginning at a dose of 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour, followed by 50 mg/kg in 500 ml 5% dextrose over four hours, and 125 mg/kg in 1000 ml 5% dextrose over 19 hours, then 150 mg/kg in 1000 ml 5% dextrose per 24 hours for an additional 48 hours. The patient will be on continuous N-acetylcysteine infusion for a total of 72 hours.
  N-acetylcysteine: Patients will be included in the trial from the onset of any hepatic coma grade and will receive NAC for the following 72 hrs.
  NAC Solutions: The N-acetylcysteine will be added to 5% dextrose in defined concentrations according to the sequence of four specific doses required for the study
  i.Solution A: 150 mg/kg bodyweight in 250 ml 5% dextrose over one hour
  ii.Solution B: 50 mg/kg in 500 ml 5% dextrose over four hours
  iii.Solution C: 125 mg/kg in 1000 ml 5% dextrose over 19 hours
  iv.Solution D: 150 mg/kg in 1000 ml 5
Arm/Group | N-acetycylcysteine | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Compare Patients Who Survive Without Transplantation to All Other Patients Enrolled in This Study (Those Who Receive a Transplant and Live, Those Who Receive a Transplant and Die, or Those Who Die Before Transplantation).
Description: The estimated minimum enrollment for any statistical validity was 100 patients. Due to low enrollment (8 participants) and the likelihood of generating any meaningful study data moving forward, the DSMB recommended the early termination of the study. Data was not collected since study was terminated.
Time Frame: 1-year follow-up
Population: Data was not collected since study was terminated, therefore there was no data to analyze.
Arm/Group | N-acetycylcysteine | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Compare Patients Who Survive Without Transplantation to All Other Patients Enrolled in This Study (Those Who Receive a Transplant and Live, Those Who Receive a Transplant and Die, or Those Who Die Before Transplantation).
Description: as for outcome 5
Time Frame: 2-year follow-up
Population: Data was not collected since study was terminated, therefore there was no data to analyze.
Arm/Group | N-acetycylcysteine | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 72-hour infusion period.
Arm/Group | N-acetycylcysteine
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetycylcysteine (N=8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination lead to zero subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No